CLINICAL TRIAL: NCT03904095
Title: Comparison Between the Analgesic Efficacy of Erector Spinae Plane Block and Psoas Compartment Block in Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sibel Seçkin Pehlivan, Teaching Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/98
Record Dates: First submitted 2019-03-28; First posted 2019-04-04 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Hip Arthropathy
Keywords: Erector spinae block; hip arthroplasty; postoperative analgesia; psoas compartment block; ultrasound
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients randomly allocated to three treatment groups: , The psoas compartment block (Group I) the ESP block group (Group II) and the control group (Group III). Blocks performed after general anesthesia induction with the Ultrasound while patients lying on surgical type at the top.
Who Masked: Participant, Investigator
Masking Description: participant care provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psoas compartment block group (PCB) (Active Comparator): Single- shot ultrasound (Esaote Mylab30) guided PCB with 15 ml 0.25% bupivacain ( Marcain 0.5%, Astra zeneca, Turkey) at the L4 vertebral level will performed preoperatively to patients in the PCB group (Group I).
  Interventions: Procedure: Psoas Compartment Block Group (GROUP I)
- Erector spinae plane block group (ESP) (Active Comparator): Single- shot ultrasound (Esaote Mylab30) guided ESP block with 15 ml 0.25% ( Marcain 0.5%, Astra zeneca, Turkey) at the L4 vertebral level will performed preoperatively to patients in the ESP group (Group II).
  Interventions: Procedure: Erector Spinae Plane block ( Group II)
- The Control group (Placebo Comparator): The Control group receive no intervention ( Group III).
  Interventions: Procedure: Control Group (GROUP III)

INTERVENTIONS:
Procedure: Psoas Compartment Block Group (GROUP I) — Psoas Compartment Block will perform preoperative to all patients in Group I. Patients in all groups will provide with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Arms: Psoas compartment block group (PCB)
Procedure: Erector Spinae Plane block ( Group II) — ESP Block will perform preoperative to all patients in ESP block group. Patients in all groups will provide with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Arms: Erector spinae plane block group (ESP)
Procedure: Control Group (GROUP III) — Control group will receive no intervention. Patients in all groups will provide with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Arms: The Control group

SUMMARY:
To evaluate the ability of Erector spina Plane block and Psoas compartment block to decrease postoperative pain and analgesia requirements in patients undergoing hip surgery.

DETAILED DESCRIPTION:
Erector spina Plane block or Psoas compartment block will performed with guided ultrasound at L4 Transverse process level would lead to adequate postoperative analgesia ,in total hip arthroplasty surgeries.

ELIGIBILITY:
Inclusion Criteria:

ASA (American Society of Anesthesiologists) I- ASA II Patients

-

Exclusion Criteria:

* history of allergy to the study medication
* refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 24 hours after surgery
  In the recovery room, all patients will given a patient- controlled analgesia device containing morphine 0.5 mg/ml, set to deliver a 1mg bolus dose of morphine with an 15 min lockout time and 6 mg 1 h limit.Total morphine consumption during the 24 hours postoperative period will recorded at 5 times intervals ( 2, 4, 6, 12, 24 hours).
Verbal analog Pain Scores on rest and movement | 24 hours after surgery
  A Research assistant, blinded to the group allocation, interviewed patients and collected data at 5 times intervals ( 2, 4, 6, 12, 24, hours) in the 24 hours postoperatively. Patients were asked to rate their pain using verbal analog scale, where 0= no pain and 10= worst pain possible.

SECONDARY OUTCOMES:
incidences of adverse effects (like nausea and vomiting) | 24 hours after surgery
  incidences of nausea and vomiting during the 24 hours postoperative period will recorded at 6 time intervals ( 2, 4, 6, 12, 24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Pehlivan, Study Director — TC Erciyes University
Locations (1):
- Sibel Seçkin Pehlivan, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel.Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Touray ST, de Leeuw MA, Zuurmond WW, Perez RS. Psoas compartment block for lower extremity surgery: a meta-analysis. Br J Anaesth. 2008 Dec;101(6):750-60. doi: 10.1093/bja/aen298. Epub 2008 Oct 22. PMID 18945717
- [Result] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Result] Tulgar S, Ermis MN, Ozer Z. Combination of lumbar erector spinae plane block and transmuscular quadratus lumborum block for surgical anaesthesia in hemiarthroplasty for femoral neck fracture. Indian J Anaesth. 2018 Oct;62(10):802-805. doi: 10.4103/ija.IJA_230_18. PMID 30443064
- See also: Related Info — http://doi.org/10.1016/j.jclinane.2018.06.033